CLINICAL TRIAL: NCT02719314
Title: Non-interventional Clinical Trial to Establish a Glucocorticoid-induced Osteoporosis Databank for Patients With Chronic Inflammatory Rheumatic Diseases or Psoriasis and Therapy With Glucocorticoids
Brief Title: Glucocorticoid-induced Osteoporosis in Patients With Chronic Inflammatory Rheumatic Diseases or Psoriasis
Acronym: Rh-GIOP
Status: Recruiting | Type: Observational
Sponsor: Prof Dr Frank Buttgereit (Other)
Responsible Party: Sponsor-Investigator, Prof Dr Frank Buttgereit, Prof Dr, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: EA1/367/14
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis; Inflammatory Rheumatism
MeSH Terms: conditions — Osteoporosis; Rheumatic Fever | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rh-GIOP(A): Glucocorticoid-induced osteoporosis (GIOP) in the context of chronic inflammatory rheumatic diseases
  Interventions: Drug: Glucocorticoid treatment
- Rh-GIOP(B): Glucocorticoid-induced osteoporosis (GIOP) in the context of psoriasis
  Interventions: Drug: Glucocorticoid treatment
- Rh-GIOP(C): Patients with or without chronic/inflammatory rheumatic diseases or psoriasis and/or without glucocorticoid treatment

INTERVENTIONS:
Drug: Glucocorticoid treatment — Glucocorticoid treatment
  Other Names: prednis(ol)one, methylprednisolone
  Groups: Rh-GIOP(A); Rh-GIOP(B)

SUMMARY:
Glucocorticoids remain to be among the most important and most frequently used anti-inflammatory and immunosuppressive or immune-modulatory acting drugs to treat rheumatic (and other) diseases. Unfortunately, glucocorticoids also exert undesired effects, especially if higher dosages have to be given over longer periods of time. The available data describing frequency and severity of these adverse effects are fragmentary. This statement is especially true for glucocorticoid-induced osteoporosis (GIOP) in the context of chronic inflammatory rheumatic diseases or (in part) psoriasis(arthritis). The state of knowledge and scientific data, being sparse, is partly conflicting and often derived from over-aged projects or studies. Therefore, there are urgent needs to work on various current questions systematically and at the highest scientific level possible. In order to address these needs, we aim at collecting and analyzing disease- and bone-related data from patients with chronic inflammatory rheumatic diseases or psoriasis and therapy with glucocorticoids, and to build a respective GIOP-Databank. Patients will attend for diagnostics, and where necessary therapy and follow-up of GIOP, according to current guidelines. Clinical, laboratory and instrumental examination results from more than 1000 patients in the first three years of the project are planned to be documented in a prospective database.

DETAILED DESCRIPTION:
Glucocorticoids remain to be among the most important and most frequently used anti-inflammatory and immunosuppressive or immune-modulatory acting drugs to treat rheumatic (and other) diseases. Unfortunately, glucocorticoids also exert undesired effects, especially if higher dosages have to be given over longer periods of time. The available data describing frequency and severity of these adverse effects are fragmentary. This statement is especially true for glucocorticoid-induced osteoporosis (GIOP) in the context of chronic inflammatory rheumatic diseases or (in part) psoriasis(arthritis), since GIOP is counted among the two most important adverse effects of glucocorticoid therapy, by both rheumatologists and patients. The state of knowledge and scientific data, being sparse, is partly conflicting and often derived from over-aged projects or studies. Therefore, there are urgent needs to work on various current questions systematically and at the highest scientific level possible. In order to address these needs, we aim at collecting and analyzing disease- and bone-related data from patients with chronic inflammatory rheumatic diseases or psoriasis and therapy with glucocorticoids, and to build a respective GIOP-Databank. Patients will attend for diagnostics, and where necessary therapy and follow-up of GIOP, according to current guidelines. Clinical, laboratory and instrumental examination results from more than 1000 patients in the first three years of the project are planned to be documented in a prospective database.

ELIGIBILITY:
Inclusion Criteria:

Every patient has to fulfill the following inclusion criteria:

* patients with (control group: without) a diagnosis of a chronic inflammatory rheumatic disease or psoriasis
* patients who (not for control groups) have/had already a glucocorticoid therapy, or patients in which the implementation of a new long-term GC therapy is expected
* patients who, according to the Dachverband Osteologie (DVO, Germany) guidelines, attend our osteoporosis and bone metabolism outpatient consultation hours or are referred by the hospital wards of the Charité for diagnosis, treatment or follow-up
* capability to understand the patient information
* consent to participation in the project and storage of data

Exclusion Criteria:

If any of the following exclusion criteria is true, the patient must not be included in this study:

* alcohol, medication and/or drug addiction
* severe psychiatric diseases limiting the comprehension of the project plan and the study protocol (persons incapable of giving informed consent)
* pregnant and lactating patients
* patients incapable of giving informed consent for any reason
* prisoners and all persons who are committed to an institution due to an official or judicial order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic inflammatory rheumatic diseases or psoriasis treated with glucocorticoids
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 2 - 5 years
  T-score (measured by DEXA; statistical evaluation on group levels, lower values are considered as being more dangerous)

SECONDARY OUTCOMES:
Mean daily glucocorticoid dosage | 1 day - 25 years
  Mean daily dosage in milligram prednisone equivalent per day (measured by questionnaire; averaged values are calculated; statistical evaluation on group levels, higher values are considered as being more dangerous)
Cumulative glucocorticoid dosage | at least 1 day - 25 years
  Cumulative glucocorticoid dosage in gram (measured by questionnaire; summed values are calculated; statistical evaluation on group levels, higher values are considered as being more dangerous)
Duration of glucocorticoid dosage | from 1 day - 25 years
  Duration of glucocorticoid therapy in days (measured by questionnaire; statistical evaluation on group levels; higher values are considered as being more dangerous)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Buttgereit, Prof Dr, Principal Investigator — Charité University Medicine Berlin (CCM)
Locations (1):
- Charité University Medicine Berlin (CCM), Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strehl C, Bijlsma JW, de Wit M, Boers M, Caeyers N, Cutolo M, Dasgupta B, Dixon WG, Geenen R, Huizinga TW, Kent A, de Thurah AL, Listing J, Mariette X, Ray DW, Scherer HU, Seror R, Spies CM, Tarp S, Wiek D, Winthrop KL, Buttgereit F. Defining conditions where long-term glucocorticoid treatment has an acceptably low level of harm to facilitate implementation of existing recommendations: viewpoints from an EULAR task force. Ann Rheum Dis. 2016 Jun;75(6):952-7. doi: 10.1136/annrheumdis-2015-208916. Epub 2016 Mar 1. PMID 26933146
- [Background] Buttgereit F. Views on glucocorticoid therapy in rheumatology: the age of convergence. Nat Rev Rheumatol. 2020 Apr;16(4):239-246. doi: 10.1038/s41584-020-0370-z. Epub 2020 Feb 19. PMID 32076129
- [Derived] Palmowski A, Boyadzhieva Z, Nielsen SM, Muche B, Hermann S, Boers M, Bliddal H, Christensen R, Wiebe E, Buttgereit F. Sex and age do not modify the association between glucocorticoids and bone mineral density in patients with rheumatoid arthritis: a cross-sectional study. Arthritis Res Ther. 2023 Jun 7;25(1):98. doi: 10.1186/s13075-023-03083-x. PMID 37287080
- [Derived] Wiebe E, Huscher D, Schaumburg D, Palmowski A, Hermann S, Buttgereit T, Biesen R, Burmester GR, Palmowski Y, Boers M, Stone JH, Dejaco C, Buttgereit F. Optimising both disease control and glucocorticoid dosing is essential for bone protection in patients with rheumatic disease. Ann Rheum Dis. 2022 Aug 11;81(9):1313-1322. doi: 10.1136/annrheumdis-2022-222339. PMID 35680387